CLINICAL TRIAL: NCT02738762
Title: Glutamine Supplementation Guided by Plasma Glutamine Levels
Brief Title: Glutamine Supplementation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: materials incomplete
Sponsor: Frisius Medisch Centrum (Other)
Responsible Party: Principal Investigator, Matty Koopmans, MSc, Frisius Medisch Centrum
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTPO 976
Record Dates: First submitted 2016-04-11; First posted 2016-04-14 (Estimated); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Glutamine; Length of Stay; Mechanical Ventilation
Keywords: intensive care; glutamine; length of stay

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Active Comparator): enteral glutamine supplementation guided by glutamine level Enteral glutamine supplementation is started (day 1) at a dose of 3 sachets per day given at 6.00, 14.00 and 22.00 hr. A sachet contains 9 grams of L-glutamine ( Glutaperos®, GLNP Life Sciences). Enteral glutamine supplementation will be given for a maximum of 10 days or until the patient is discharged from the ICU
  Interventions: Other: glutamine supplementation
- control group (No Intervention): patients receive normal treatment, no glutamine supplementation

INTERVENTIONS:
Other: glutamine supplementation — glutamine supplementation guided by glutamine levels in plasma
  Arms: intervention group

SUMMARY:
Earlier studies showed a benefit in survival when glutamine was given intravenously and these studies lead to recommendations that glutamine should be given to critically ill patients. The ESPEN guidelines recommend 0,2-0,4 g/kg/d intravenous glutamine added to standard parenteral nutrition .

Until recently it was not possible to obtain a plasma glutamine level fast enough to consider the result for clinical decision making. With the availability of a Point of Care (POCT) measurement of plasma glutamine level a measurement can be performed short after the collection of blood. This offers the possibility to identify a patient with a low plasma glutamine level shortly after admission and use repeated measurements for evaluation of the response to supplementation of glutamine.

DETAILED DESCRIPTION:
* At admission (day 0) a plasma glutamine level is measured. The measurement can be performed from blood taken for the first arterial blood gas analysis. Patients are eligible for the study when the plasma glutamine level is lower than 420 µmol/l.
* After informed consent is obtained patients are randomised to receive enteral glutamine or not ( the control group). Enteral glutamine supplementation is started (day 1) at a dose of 3 sachets per day given at 6.00, 14.00 and 22.00 hr. A sachet contains 9 grams of L-glutamine ( Glutaperos®, GLNP Life Sciences).
* Enteral glutamine supplementation will be given for a maximum of 10 days or until the patient is discharged from the ICU.
* Plasma glutamine levels will be measured four times a day, at 06.00, 12.00, 18.00 and 00.00 hours, concurrently with the standard arterial blood gas analyses so no extra blood is taken from the patient.
* On day 3 at 12.00 hours the dose of glutamine will be increased to 3 times 2 sachets if plasma glutamine level is still below 420 µmol/l.
* From day 3 ( 12.00 hrs) until day 10 ( end of study) the dosage of enteral glutamine will be evaluated daily at 12.00 hours. When the plasma glutamine level is higher than 420 µmol/l the dosage of enteral glutamine will be adjusted according to the schedule below.
* In patients who randomized to the control group, the plasma glutamine level will be measured daily at 12.00 hr concurrently with standard arterial blood gas analysis

ELIGIBILITY:
Inclusion Criteria:

* all patients admitted to the ICU with an expected stay of 48 hours or longer
* glutamine level lower thand 420 mmol/l

Exclusion Criteria:

* age under 18 years
* readmission to the ICU
* contra indication for enteral nutrition
* use of total parental nutrition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
amount of enteral glutamine supplementation glutamine level | 10 days
  amount of enteral glutamine supplementation needed to increase the plasma
length of mechanical ventilation | 10 days
  difference in length of mechanical ventilation between two groups

SECONDARY OUTCOMES:
hospital mortality | 6 months
  difference in hospital mortality between two groups

CONTACTS AND LOCATIONS:
Overall Officials: Matty Koopmans, MSc, Principal Investigator — MCL

IPD SHARING:
Plan to Share IPD: No
patient data is anonym